CLINICAL TRIAL: NCT00804830
Title: Phase 2 Study With Avastin and Doxorubicin Postoperatively for Patients With Anaplastic Thyroid Cancer
Brief Title: Avastin and Doxorubicin Postoperatively for Patients With Anaplastic Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of response
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-001783-75
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Thyroid Neoplasms; Carcinoma; Thyroid Cancer; Metastatic Cancer
Keywords: adjuvant; Anaplastic thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma; Neoplasm Metastasis; Thyroid Carcinoma, Anaplastic | interventions — Bevacizumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy (Experimental): Treatment with Avastin 15 mg/kg q3w and doxorubicin 20 mg q1w for 6 months.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Avastin 15 mg/kg q3w and doxorubicin 20 mg q1w
  Other Names: Avastin 15 mg/kg q3w and doxorubicin 20 mg q1w

SUMMARY:
Anaplastic Thyroid Cancer is a very aggressive disease. The investigators believe that angiogenesis is very important for these tumors to progress. Preclinical data is suggesting this. This is why we we prospectively want to treat these patients with avastin (and doxorubicin). However, local control is of major concern. Therefore, patients are initially treated with hyperfractionated radiotherapy and undergo surgery. Then they can enter this study.

DETAILED DESCRIPTION:
Patients with Anaplastic Thyroid Cancer have a poor prognosis. We will treat the patients initially with our standard radiochemotherapy, which consists of doxorubicin 20mg fixed dose/week and hyperfractionated radiotherapy 1,6 Gy twice daily up to 46 Gy in total. The first week during radiotherapy, they will also receive Avastin 15mg/kg. 1-2 weeks after radiotherapy patients will undergo surgery of their primary tumor. After this "standard" therapy patients can be included in this study. Treatment is 20 mg fixed dose doxorubicin q1w and avastin 15mg/kg q3w. Treatment will continue maximum 6 months or until progress or until intolerable side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* cytologically or histologically verified anaplastic thyroid cancer
* completed standard therapy
* operated with R0 or R1 surgery
* Performance Status 0-2 (if pulmonary mets PS 0-1)
* normal wound healing
* neutrophils > 1,5 million/ml
* platelets > 100 million/ml
* bilirubin < 2 ULN
* creatinin < 150mikromol/L

Exclusion Criteria:

* PS 3-4 (if pulmonary mets 2-4)
* R2 resection of primary tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2-5 years

SECONDARY OUTCOMES:
Response rate | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tennvall, MD, PhD, Principal Investigator — Dep of Oncology, Lund University Hospital
Locations (3):
- Sweden (3):
  - Jubileumskliniken, Sahlgrenska universitetsjukhuset, Gothenburg
  - Dep of Oncology, Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm